CLINICAL TRIAL: NCT03098342
Title: Comparison of Efficacy and Safety Between Methylene Blue-mediated Photodynamic Therapy and 5% Amorolfine Nail Lacquer for Toenail Onychomycosis Treatment in Asians
Brief Title: Comparison of Efficacy and Safety Between Methylene Blue-mediated Photodynamic Therapy and 5% Amorolfine Nail Lacquer for Toenail Onychomycosis Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chulalongkorn University (Other)
Collaborators: King Chulalongkorn Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CU_MBPDT_for_Onychomycosis
Record Dates: First submitted 2017-02-20; First posted 2017-03-31 (Actual); Last update posted 2017-03-31 (Actual); Status verified 2017-02

CONDITIONS: Onychomycosis of Toenail
Keywords: Onychomycosis; photodynamic therapy; methylene blue; amorolfine, nail lacquer; Asians
MeSH Terms: conditions — Onychomycosis | interventions — Methylene Blue; amorolfine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MB-PDT for Onychomycosis (Experimental)
  Interventions: Procedure: Methylene blue-mediated photodynamic therapy
- Amorolfine for Onychomycosis (Active Comparator)
  Interventions: Drug: Amorolfine 5% Nail Lacquer

INTERVENTIONS:
Procedure: Methylene blue-mediated photodynamic therapy — Using the 2% MB aqueous solution as a photosensitiser. After the rest period, the lesion was immediately illuminated with incoherent red light (peak emission spectrum at 630-640 nm)
  Other Names: Incoherent red light (peak emission spectrum at 630-640 nm); Methylene blue
  Arms: MB-PDT for Onychomycosis
Drug: Amorolfine 5% Nail Lacquer — Patients will be detailed instruction regarding the use of 5% Amorofine Nail Lacquer (Loceryl®) as its recommended protocol.
  Arms: Amorolfine for Onychomycosis

SUMMARY:
Study centre and address

King Chulalongkorn Memorial Hospital

Primary objective

To compare the efficacy and the safety of methylene blue-mediated photodynamic therapy and 5% amorolfine nail lacquer for toenail onychomycosis in Asians

DETAILED DESCRIPTION:
• Research Design

Randomized, single-blind clinical trial

• Research Methodology

Target population

* 42 Patients, aged between 18-90 years old, with distal and lateral subungual toenail onychomycosis diagnosed clinically and mycologically
* Patients were recruited from Dermatology clinic, King Chulalongkorn Memorial Hospital

  * Exclusion criteria

    1. Those with nail changes because of skin disease or associated systemic diseases
    2. Those who had previously used anti-fungal medications within 3 months for systemic and 1 month for topical therapy.
  * Methods

    1. Patients will be informed of the details of the study including predicted possible adverse events due to the treatments and primary aids.
    2. They will be included in stratified randomly by poor prognostic factors, then divided into two groups (A: methylene blue-mediated photodynamic therapy (MB-PDT) and B: 5% Amorolfine Nail Lacquer by block randomization of size 4 and 6.
    3. For 24 weeks,
* Group A

  * The use of PDT consisting of 6 treatment sessions with interval of 15 days between each session
  * Patient will be instructed that apply 40% urea cream under occlusive dressing for 5 days prior to PDT.
* Group B

  * Patients will be detailed instruction regarding the use of 5% Amorolfine Nail Lacquer as its recommended protocol.
  * Total duration of the follow-up is 18 months

Evaluation tool

* Nail photographs by using dermoscope for onychomycosis severity index (OSI) evaluation
* Either Scrape or nail clipping, which is positive prior to the treatment, will be performed for microscopic study and culture.
* Safety will be assessed through adverse events.
* Patients' satisfaction will be evaluated at the end of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients, aged between 18-90 years old, with distal and lateral subungual toenail onychomycosis diagnosed clinically and mycologically

  * Clinical signs of onychomycosis as following:

    * Discoloration
    * Dystrophy of nail plate
    * Subungual hyperkeratosis
    * Onycholysis
  * Confirmed by:

    * Positive culture of dermatophyte or non-dermatophyte (must be isolated from sequential specimens) and/or
    * Positive microscopic evidence*
  * *any of these methods, direct microscopy (KOH preparation), nail plate culture on Sabouraud's dextrose agar (SDA), histopathological examination of nail clippings using PAS staining (HPE-PAS), histopathological examination of nail clippings using GMS staining (HPE-GMS), polymerase chain reaction

Exclusion Criteria:

* Those with nail changes because of skin disease or associated systemic diseases
* Pregnancy or lactating woman
* Those who are allergic to amorolfine, methylene blue
* Those who are photosensitive to visible light
* Those who had previously used anti-fungal medications within 3 months for systemic and 1 month for topical therapy.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2017-06-01 (Estimated); Primary Completion 2018-12-30 (Estimated); Study Completion 2019-01-31 (Estimated)

PRIMARY OUTCOMES:
Onychomycosis severity index (OSI) | Change from baseline Onychomycosis severity index at every 2 weeks through the MB-PDT treatment completion, 12 weeks; then change from baseline Onychomycosis severity index at every 8 weeks through the study completion, an average of 18 months.
  Photographs taken by using a dermoscope were evaluated by two independent dermatologists.

CONTACTS AND LOCATIONS:
Overall Officials: Natthamon Bowornsathitchai, MD, Principal Investigator — Chulalongkorn University
Locations (1):
- King Chulalongkorn Memorial Hospital, Bangkok, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided